CLINICAL TRIAL: NCT05050994
Title: Ultrasound Guided Partial Microwave Ablation of the Spleen Due to Secondary Splenomegaly in Children - a Study of Feasibility and Acceptability
Brief Title: Ultrasound Guided Microwave Ablation of Splenomegaly in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Thomas Casswall, Clinical Professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-06155
Record Dates: First submitted 2021-09-10; First posted 2021-09-21 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-09

CONDITIONS: Splenomegaly; Congestive, Chronic; Panhematopenia; Splenic; Portal Hypertension
Keywords: Microwave ablation
MeSH Terms: conditions — Splenomegaly; Bronchiolitis Obliterans Syndrome; Hypertension, Portal

STUDY DESIGN:
Intervention Model Description: Prospective observational pilot trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Microwave ablation (Experimental): Patients receiving microwave ablation of splenomegaly
  Interventions: Procedure: Microwave ablation

INTERVENTIONS:
Procedure: Microwave ablation — Children with symptomatic secondary splenomegaly will receive partial microwave ablation of spleen (up to 40-50% of total volume)

SUMMARY:
Children with liver cirrhosis frequently develops portal hypertension. One of the serious complications to portal hypertension is splenomegaly, which may result in pancytopenia, especially thrombocytopenia that may cause bleeding tendencies.

Symptomatic splenomegaly is often treated with partial splenic embolization (PSE). PSE is effective but may give rise to postembolization syndrome not well tolerated in the pediatric population. In adults, microwave ablation (MWA) has been used to treat splenomegaly with promising results but with less post-operative pain. Our study is a pilot trial to evaluate the feasibility and acceptability of this treatment in children.

DETAILED DESCRIPTION:
The ablation will be performed under general anesthesia by an experienced interventional radiologist. Ultrasound will be used for peri-operative assessment and the microwave antenna will be inserted under ultrasound guidance focusing on the middle to inferior part of the spleen to avoid harm to the diaphragm. After the emission of microwaves for up to 5 minutes, the antenna will be pulled back and the emission will be repeated until the ablation zone is approximately 1 cm from the splenic surface. In this way, two or three overlapping areas will be ablated with every insertion of the antenna. The ablation zones will be visible as hyperechoic areas on b-mode ultrasound during operation, and the goal is to ablate up to 40-50% of the total volume of the spleen (as estimated by the radiologist). If the ablated volume is less than 40-50% at follow up, the procedure can be repeated in a second session for additional effect.

ELIGIBILITY:
Inclusion Criteria:

* Spleen length > +2 standard deviations of normal limit
* Platelet count below 30-35 x 109 cells/L and a history of bleeding tendencies
* Symptoms of portal hypertension such as splenomegaly, thrombocytopenia, leucopenia, ascites, esophageal or gastric varices, hypertensive gastropathy, anal hemorrhoids and increased portal scintigraphy index, where alternative methods have not been enough or suitable
* A necessity for reduction of splenic volume due to splenic inhibition of motion and activity in the child

Exclusion Criteria:

* Age younger than 10 or older than 17 years of age
* Legal guardians or child do not give consent
* Ongoing infection

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Platelet count | Base line and 1, 3, 6 and 12 months follow up
  Difference between platelet count before MWA and at 1, 3, 6 and 12 months after treatment

SECONDARY OUTCOMES:
Number of MWA | Within 12 months
  Number of MWA to achieve goal with platelet count > 50 x 109 cells/L or reducing functional spleen with 50%
Effect on blood cell count | Base line and 1, 3, 6 and 12 months follow up
  Effect on red and white blood cell count
Effect on liver function | Base line and 1, 3, 6 and 12 months follow up
  Measurement of AST, ALT, ALP, GGT, bilirubin, cholinesterase, albumin, ammonia
Effect on coagulation | Base line and 1, 3, 6 and 12 months follow up
  Measurement of PT-INR, APTT, D-dimer, fibrinogen, ROTEM with fibrinogen, antithrombin, von Willebrand activity (vWGP1bA), factor VIII enzyme
Maximal pain | Day of surgury and the following 7 days
  Measured using the Visual Analog Scale, a numerical rating scale from 0 - 10 where 0 is no pain and 10 is worst imaginable pain.
Use of analgesic drugs | Day of surgury and the following 7 days
  The administration of standardized analgesic drugs will be recorded
Days of hospitalization | 1 month
  How many days the patient stays in hospital after ablation
Acceptability of treatment | 1 month after ablation
  Measured as parents preferred future treatment and as if the method could be recommended to a family with a child with a similar medical condition

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Casswell, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden